CLINICAL TRIAL: NCT00904540
Title: Open-Label Study Assessing the Efficacy of Topical Lidocaine Patch in Treatment of Low Back Pain
Brief Title: Topical Lidocaine Patch in Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr Director, Clinical R & D, Endo Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3220-006
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Acute and Chronic Non-radicular LBP
MeSH Terms: interventions — Lidoderm

ARMS (1):
- Lidoderm® (Experimental): Commercially available Lidoderm (lidocaine patch 5%), up to four patches applied topically once daily (q24h) to the area of maximal peripheral pain
  Interventions: Drug: Lidoderm®

INTERVENTIONS:
Drug: Lidoderm® — Patients participated in a 6-week treatment period. Commercially available Lidoderm (lidocaine patch 5%) was provided to patients with up to four patches applied topically once daily (q24h) to the area of maximal peripheral pain. Patients were stratified into the following groups at enrollment: acute (<6 weeks) LBP, subacute (6 weeks to <3 months) LBP, short-term chronic (3 months to 12 months, inclusive) LBP, and long-term chronic (>12 months LBP)
  Other Names: Lidocaine patch 5%

SUMMARY:
Patients with acute or chronic Lower Back Pain (LBP) participated in a Phase IV clinical trial to assess the effectiveness of Lidoderm administered once daily (q24h) for 2 weeks in the treatment of acute and chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* Non-radicular LBP pain for

  ≤12 months (non-radicular defined as LBP that does not radiate below the mid-buttock and with no sensory symptoms in the leg)
* Had LBP as the primary source of pain. Patients may have had mild to moderate spinal stenosis and no radicular symptoms
* Had an average daily pain intensity score of >4 on a 0 to 10 scale, with 0 being no pain and 10 being pain as bad as the patients have ever imagined (Question 5 of BPI) within 24 hours prior to the screening visit.
* Had a normal neurological examination, including:

  * Motor strength
  * Sensory testing (light touch, pinprick, and vibration)
  * Deep tendon reflexes

Patients were eligible for participation in the long-term chronic (>12 months) group of the study if they also:

* Had LBP for greater than one year. Patients may have had any of the following: lumbar degenerative disc disease, internal disc disruption, mild-to-severe spinal stenosis, degenerative scoliosis and spondylolisthesis, facet arthropathy

Exclusion Criteria:

* Had a history of greater than one back surgery or one back surgery within 3 months of study entry
* Had severe spinal stenosis and radicular symptoms
* Had any other chronic pain condition that, in the opinion of the investigator, would have interfered with patient assessment of LBP relief
* Had received an epidural steroid/local anesthetic injection within 2 weeks prior to study entry
* Had received trigger point injections within 2 weeks prior to study entry
* Had received Botox Injections within 3 months prior to study entry
* Were taking a lidocaine-containing product that could not be discontinued while receiving Lidoderm
* Were taking class 1 anti-arrhythmic drugs (e.g., mexiletine, tocainide)

Patients were excluded from participation in the long-term chronic (>12 months) group if they also:

* Had an undefined spinal diagnosis
* Had a history of lumbar spine surgery within 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2002-03; Primary Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Mean change in average daily intensity (Question 5 of Brief Pain Inventory [BPI] Questionnaire) from baseline to Week 2 | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 14), V5 (Day 28), V6/EOS (Day 42)

SECONDARY OUTCOMES:
Mean change from baseline to Week 6 in average pain intensity (Question 5 of the BPI) | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 14), V5 (Day 28), V6/EOS (Day 42)
Mean change from baseline to Week 2 and to Week 6 in Neuropathic Pain Scale (NPS) composite scores | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 14), V5 (Day 28), V6/EOS (Day 42)
QOL: change from baseline to Week 2 to Week 6 in Question 9 of the BPI, in Beck Depression Inventory Questionnaire, and the Patient and Investigator Global Assessment of Patch Satisfaction and Pain Relief | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 14), V5 (Day 28), V6/EOS (Day 42)
Safety assessments include AEs, clinical laboratory tests, vital signs, physical/neurological examinations, and dermal/sensory assessments. | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 14), V5 (Day 28), V6/EOS (Day 42)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals
Locations (7):
- United States (7):
  - Phoenix, Arizona
  - Mill Valley, California
  - Weston, Florida
  - Bethpage, New York
  - Charlotte, North Carolina
  - Allentown, Pennsylvania
  - Madison, Wisconsin